CLINICAL TRIAL: NCT00139256
Title: Randomized Controlled Trial of Antepartum Betamethasone Treatment for Prevention of Respiratory Distress in Infants Born by Elective Cesarean Section
Brief Title: Antepartum Betamethasone Treatment for Prevention of Respiratory Distress in Infants Born by Elective Cesarean Section
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow enrollment and lack of funds.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lucky Jain, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0894-2003
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Glucocorticoid; Antepartum Betamethasone Treatment; Elective Cesarean Section; Respiratory Distress in Infants
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Betamethasone (Experimental): Betamethasone injection
  Interventions: Drug: Betamethasone
- Placebo (Placebo Comparator): Placebo injection
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: Betamethasone — Betamethasone injection

SUMMARY:
This is a randomized, multicenter, double blind, placebo controlled trial of betamethasone versus a placebo given prior to the mothers at term and near term gestation (>34 and <40 weeks of gestation) who are scheduled to undergo a planned Cesarean section. The study design is to determine the efficacy and safety of betamethasone in the prevention of breathing problems commonly seen in this population.

In infants born by elective Cesarean section, it is hypothesized that antenatal betamethasone treatment will reduce the risk of neonatal intensive care unit (NICU) admission from 11% to 8% and/or oxygen therapy +/- positive pressure ventilation (PPV) for >30 minutes from 4.5% to 2.5%.

DETAILED DESCRIPTION:
The purpose of this pilot study is to determine if antepartum betamethasone given to mothers undergoing elective cesarean section (ECS) delivery at term or near term gestation (>34 and < 40 weeks of gestation) is safe and feasible in reducing neonatal respiratory morbidity and the related admissions to neonatal intensive care units (NICU).

The data from this pilot study will be used to support a NIH application for a multicenter randomized trial to determine, if compared to placebo treatment, antenatal betamethasone initiated 2-7 days prior to an ECS results in decreased occurrence of respiratory morbidity and NICU admissions in the newborn.

The multicenter protocol was recently reviewed by the NICHD network for clinical trial. The reviewers were enthusiastic about the scientific merit and public health importance of the study but asked for a pilot study to determine feasibility before launching the national trial. Given the rise in the rate of CS deliveries, we project substantial health cost savings from this preventive strategy if it were found to be successful in reducing neonatal morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women >/= 34 weeks gestation scheduled to undergo operative delivery within 48-72 hours after study enrollment

Exclusion Criteria:

* Known contraindication to the use of betamethasone in the mother
* Known lethal or non-lethal congenital anomaly diagnosed antenatally
* Spontaneous labor
* Premature rupture of membranes

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-08; Primary Completion 2007-04 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome to be studied is the need for NICU admission and/or oxygen therapy or PPV for >30 minutes. | 24 hours
  Respiratory distress in the first 24 hours after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Lucky Jain, M.D., Principal Investigator — Emory University Department of Pediatrics, Division of Neonatology
Locations (1):
- Emory University affiliated newborn intensive care units, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Sotiriadis A, McGoldrick E, Makrydimas G, Papatheodorou S, Ioannidis JP, Stewart F, Parker R. Antenatal corticosteroids prior to planned caesarean at term for improving neonatal outcomes. Cochrane Database Syst Rev. 2021 Dec 22;12(12):CD006614. doi: 10.1002/14651858.CD006614.pub4. PMID 34935127